CLINICAL TRIAL: NCT03426033
Title: Phase 1, Drug-Drug Interaction Study To Evaluate The Effect Of Multiple Doses Of ISIS 681257 40 mg Subcutaneous Injections On The Pharmacokinetics And Pharmacodynamics Of Warfarin In Healthy Subjects
Brief Title: Drug-drug Interaction Study to Evaluate the Effect of ISIS 681257 on Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akcea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ISIS 681257-CS10
Record Dates: First submitted 2018-01-03; First posted 2018-02-08 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Elevated Lipoprotein(a); Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Warfarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single dose of warfarin (Experimental): Single dose of warfarin administered to obtain pharmacokinetic information.
  Interventions: Drug: Warfarin
- Warfarin in combination with ISIS 681257 (Experimental): ISIS 681257 administered and pharmacokinetic assessments are taken. Then ISIS 681257 is administered with warfarin and additional pharmacokinetic information is obtained.
  Interventions: Drug: ISIS 681257; Drug: Warfarin

INTERVENTIONS:
Drug: ISIS 681257 — Xmg dose administered as a subcutaneous injection
  Arms: Warfarin in combination with ISIS 681257
Drug: Warfarin — 25mg tablet administered orally

SUMMARY:
This is a single center, open label, single sequence, two-treatment, two-period drug-drug interaction study to evaluate the effect of multiple doses of ISIS 681257 on the pharmacokinetics of a single dose of warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Motivated and available for duration of study and willing to adhere to protocol
* Males who are unable to procreate or agree to contraception throughout study
* Females who are postmenopausal or surgically sterile
* BMI between 18.5 and 30 kg/m2
* Weighing greater than or equal to 50kg
* Normal lab results
* No known diseases or significant findings on physical exam

Exclusion Criteria:

* Females of childbearing potential
* Reactions/infection at injection site
* Hypersensitivity to any drugs or similar drugs to those used in the study
* Conditions or disease that may interfere with study drug
* Any significant diseases
* Known history or familial history of bleeding disorders
* Drug dependency or abuse
* Illness within 28 days
* Previous exposure to other investigational drug within 28 days
* Blood donations within 28 days

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-02-25 (Actual); Study Completion 2018-02-25 (Actual)

PRIMARY OUTCOMES:
The plasma concentrations of warfarin and ISIS 681257 will be measured at each individual time point. | Each day for days 1-10 and 15-45
  To evaluate the effect of multiple doses of ISIS 681257 40 mg subcutaneous injections on the pharmacokinetics of a single oral dose of warfarin in healthy adult subjects.

SECONDARY OUTCOMES:
The safety of ISIS 681257 by the incidence of treatment-emergent adverse events. | 45 days
  To evaluate the safety and tolerability of multiple doses of ISIS 681257 40 mg subcutaneous injections when coadministered with a single oral dose of warfarin in healthy adult subjects.
Prothrombin Time will be measured by testing blood samples at each individual time point. | Each day for days 1-7 and 15-21
  To evaluate the effect of multiple doses of ISIS 681257 40 mg subcutaneous injections on the pharmacodynamics (anticoagulant activity) of a single oral dose of warfarin in healthy adult subjects.
International normalized ratio will be measured at each individual time point by comparing prothrombin time to the normal mean prothrombin time. | Each day for days 1-7 and 15-21
  To evaluate the effect of multiple doses of ISIS 681257 40 mg subcutaneous injections on the pharmacodynamics (anticoagulant activity) of a single oral dose of warfarin in healthy adult subjects.
Activated partial thromboplastin time will be measured by testing blood samples at each individual time point. | Each day for days 1-7 and 15-21
  To evaluate the effect of multiple doses of ISIS 681257 40 mg subcutaneous injections on the pharmacodynamics (anticoagulant activity) of a single oral dose of warfarin in healthy adult subjects.
The plasma concentrations of warfarin and ISIS 681257 will be measured at each individual time point. | Each day for days 1-10 and 15-45
  To evaluate the effect of a single dose of warfarin on the pharmacokinetics of a single subcutaneous 40 mg injection of ISIS 681257 in healthy adult subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Site, Mount Royal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Milosavljevic MN, Stefanovic SM, Pejcic AV. Potential Novel RNA-Targeting Agents for Effective Lipoprotein(a) Lowering: A Systematic Assessment of the Evidence From Completed and Ongoing Developmental Clinical Trials. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):1-12. doi: 10.1097/FJC.0000000000001429. PMID 37070852